CLINICAL TRIAL: NCT05503953
Title: A Multicenter, Randomized, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of AGSAVI in Patients With Essential Hypertension Inadequately Controlled With AGLS
Brief Title: Phase III Study to Evaluate the Efficacy and Safety of AGSAVI in Patients With Essential Hypertension Inadequately Controlled With AGLS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Collaborators: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG-1705_P3
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGSAVI (Experimental)
  Interventions: Drug: AGSAVI
- AGLS (Active Comparator)
  Interventions: Drug: AGLS

INTERVENTIONS:
Drug: AGSAVI — Uptitation
  Arms: AGSAVI
Drug: AGLS — Uptitration
  Arms: AGLS

SUMMARY:
A multicenter, Randomized, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of AGSAVI in Patients with Essential Hypertension Inadequately Controlled with AGLS

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patient who satisfied below condition at Visit 1.

  * patient who takes antihypertensive drug

    * 140mmHg <= MSSBP < 200mmHg
    * 130mmHg <= MSSBP < 200mmHg at or before visit 1(In high-risk patients)
  * patient who doesn't take antihypertensive drug

    * 160mmHg <= MSSBP < 200mmHg
* Hypertension patient who satisfied below condition at Visit 2.

  * 140mmHg <= MSSBP < 200mmHg at Visit 2
  * 130mmHg <= MSSBP < 200mmHg at or before Visit 1(In high-risk patients)

Exclusion Criteria:

* Patient who have received 4 or more antihypertensive drug
* Patient with 20mmHg>= of difference in MSSBP or 10mmHg>= of difference in MSDBP between 2 times of BP measuring at Visit 1
* Patient with MSDBP >= 120mmHg at Visit 1 or 2
* Patient with secondary hypertension(including past medical history)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2022-09-05 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of MSSBP(Mean Sitting Systolic Blood Pressure) | From Baseline(Visit 2) to Visit 5(For 10 weeks)
  Change of MSSBP(Mean Sitting Systolic Blood Pressure) From Baseline to Visit 5(For 10 weeks)